CLINICAL TRIAL: NCT01566721
Title: A Phase III Prospective, Two-Cohort Non-Randomized, Multi-Centre, Multinational, Open-Label Study to Assess the Safety of Assisted- and Self-Administered Subcutaneous Trastuzumab as Therapy in Patients With Operable HER2-Positive Early Breast Cancer
Brief Title: A Safety and Tolerability Study of Assisted and Self-Administered Subcutaneous (SC) Herceptin (Trastuzumab) as Adjuvant Therapy in Early Human Epidermal Growth Factor Receptor 2 (HER2)-Positive Breast Cancer
Acronym: SafeHER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MO28048; 2011-005328-17 (EudraCT Number)
Record Dates: First submitted 2012-03-22; First posted 2012-03-29 (Estimated); Results first posted 2017-04-18 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort A: SC Herceptin by Needle/Syringe (Experimental): Participants will receive SC Herceptin by an assisted administration using a conventional syringe and needle/vial formulation.
  Interventions: Drug: Herceptin
- Cohort B: SC Herceptin by SID (Experimental): Participants will receive SC Herceptin with assisted and/or self-administered use of an SID. The first administration will be performed by a trained healthcare professional. If well tolerated and the participant is willing and judged competent to perform self-administration, subsequent administration of SC Herceptin may be performed by the participant.
  Interventions: Drug: Herceptin

INTERVENTIONS:
Drug: Herceptin — Herceptin will be given as 600 mg SC (into thigh) on Day 1 of each 3-week cycle for up to 18 cycles.
  Other Names: Trastuzumab

SUMMARY:
This multicenter, two-cohort, non-randomized, open-label study will evaluate the safety and tolerability of assisted and self-administered SC Herceptin as adjuvant therapy in participants with early HER2-positive breast cancer following tumor excision. Participants will receive Herceptin 600 milligrams (mg) SC every 3 weeks for 18 cycles, either by an assisted administration using a conventional syringe and needle/vial formulation (Cohort A) or with assisted and self-administration using a single-use injection device (SID) in selected participants (Cohort B).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed early invasive HER2-positive carcinoma of the breast with no evidence of residual, locally recurrent, or metastatic disease and defined as clinical Stage I to IIIC that is eligible for treatment with Herceptin
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Screening left ventricular ejection fraction (LVEF) greater than or equal to (≥) 55%

Exclusion Criteria:

* Previous neoadjuvant or adjuvant breast cancer treatment with an approved or investigational anti-HER2 agent
* History of other malignancy except for curatively treated carcinoma in situ of the cervix, basal cell carcinoma, or curatively treated malignancies (other than breast cancer) where the participant has been disease-free for at least 5 years
* Past history of ductal carcinoma in situ treated with any systemic therapy or with radiation therapy to the ipsilateral breast where invasive cancer subsequently developed
* Metastatic disease
* Inadequate bone marrow, hepatic, or renal function
* Serious cardiac or cardiovascular disease including uncontrolled hypertension or history of hypertensive crisis or hypertensive encephalopathy
* History of severe allergic or immunological reactions, such as difficult-to-control asthma
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2577 (Actual)
Dates: Start 2012-05-17 (Actual); Primary Completion 2015-03-10 (Actual); Study Completion 2020-02-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (437):
- University "Mother Theresa" Hospital Center; Oncology Department, Tirana, Albania
- CPMC; Service d'Oncologie Médicale, Algiers, Algeria
- Argentina (3):
  - Fundación CENIT para la Investigación en Neurociencias, Buenos Aires
  - Hospital Britanico; Oncologia, Buenos Aires
  - Instituto De Investigaciones Clinicas Zarate, Zárate
- Australia (9):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - St George Hospital; Cancer Care Centre, Kogarah, New South Wales
  - Prince of Wales Hospital; Oncology, Randwick, New South Wales
  - Princess Alexandra Hospital; Division of Cancer Services, Woolloongabba, Queensland
  - Queen Elizabeth Hospital; Medical Oncology, Woodville South, South Australia
  - Western Hospital, Footscray, Victoria
  - Peninsula and South Eastern Haematology and Oncology Group, Frankston, Victoria
  - Cabrini Medical Centre; Oncology, Malvern, Victoria
  - Royal Perth Hospital; Department of Medical Oncology, Perth, Western Australia
- Bosnia and Herzegovina (2):
  - University Clinical Center of the Republic of Srpska, Banja Luka
  - Clinic of Oncology, University Clinical Center Sarajevo, Sarajevo
- Brazil (6):
  - Hospital Sao Rafael - HSR, Salvador, Estado de Bahia
  - Centro de Oncologia da Bahia - CENOB, Salvador, Estado de Bahia
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Hospital Perola Byington, São Paulo, São Paulo
- Bulgaria (3):
  - Complex Oncology Center - Plovdiv First Internal Chemotherapy Department, Plovdiv
  - MHAT Serdika; Department of medical oncology, Sofia
  - SHATOD - Sofia, Sofia
- Canada (8):
  - Cross Cancer Institute ; Dept of Medical Oncology, Edmonton, Alberta
  - British Columbia Cancer Agency (Bcca) - Vancouver Cancer Centre, Vancouver, British Columbia
  - The Moncton Hospital, Moncton, New Brunswick
  - Lakeridge Health Oshawa; Oncology, Oshawa, Ontario
  - St. Michael'S Hospital, Toronto, Ontario
  - Windsor Regional Cancer Centre, Windsor, Ontario
  - CSSS champlain - Charles-Le Moyne, Greenfield Park, Quebec
  - Mcgill University - Royal Victoria Hospital; Oncology, Montreal, Quebec
- Chile (4):
  - Centro Oncológico Antofagasta, Antofagasta
  - Instituto Nacional del Cancer, Santiago
  - Sociedad de Investigaciones Medicas Ltda (SIM), Temuco
  - Hospital Carlos Van Buren, Servicio de Oncologia, Valparaíso
- Colombia (2):
  - Clinica del Country, Bogotá
  - Clínica Imbanaco; Oncology, Cali
- Croatia (2):
  - Clinical Hospital Osijek; Dept For Oncology & Radiotherapy, Osijek
  - Clinical Hospital Centre Zagreb, Zagreb
- Czechia (3):
  - Masarykův onkologický ústav; Klinika komplexní onkologické péče, Brno
  - Fakultní nemocnice Olomouc, Olomouc
  - Fakultní Nemocnice V Motole; Radioterapeuticko-Onkologicke Oddeleni, Prague
- Hospital Metropolitano de Santiago, Santiago de los Caballeros, Dominican Republic
- Ecuador (3):
  - Instituto de Cáncer SOLCA Cuenca; Oncología, Cuenca
  - Solca Guayaquil- Sociedad de Lucha Contra El Cáncer; Oncology, Guayaquil
  - Hospital Solca Quito; Oncologia, Quito
- Egypt (3):
  - Alexandria Uni ; Medical Oncology, Alexandria
  - Manial Specialized Hospital; Oncology, Cairo
  - Nci; Oncology Dept, Cairo
- Hospital Oncologia; Oncology, San Salvador, El Salvador
- France (45):
  - HOPITAL JEAN MINJOZ; Oncologie, Besançon
  - Clinique Tivoli; Sce Radiotherapie, Bordeaux
  - Polyclinique Bordeaux Nord Aquitaine; Chimiotherapie Radiotherapie, Bordeaux
  - Ch De Fleyriat; Pneumologie 1, Bourg-en-Bresse
  - Hopital Augustin Morvan; Federation De Cancerologie, Brest
  - Ch De Brive La Gaillarde; Radiotherapie Oncologie, Brive-la-Gaillarde
  - Clinique Sainte Marie; Chimiotherapie, Chalon-sur-Saône
  - Fondation Clement Drevon; Oncology, Dijon
  - Centre Georges-François Lecler; Ctr de Lutte Contre le Canc, Dijon
  - Ch De La Dracenie; Hopital De Jour, Draguignan
  - Hopital Prive Drome Ardeche; Chir 2A 2B, Guilherand-Granges
  - Clinique Sainte Marguerite; Oncologie Medicale, Hyères
  - CHD Les Oudairies, La Roche-sur-Yon
  - Hopital Albert Michallon; Oncologie, La Tronche
  - Ch Du Mans; Medecine Hematologie Oncologie, Le Mans
  - Clinique Victor Hugo, LeMans
  - Centre Hartmann, Levallois-Perret
  - Polyclinique Du Bois; Centre Bourgogne, Lille
  - Hopital Claude Huriez; Medecine Interne Oncologie, Lille
  - Ch Bretagne Sud Site Scorff; Oncologie Medicale, Lorient
  - CH Bretagne Sud Site Bodelio; Oncologie Radiotherapie, Lorient
  - Ctre Consultations La Sauvegarde, Lyon
  - Hôpital Saint Joseph; Oncologie Medicale, Marseille
  - Hopital Clinique Claude Bernard; Oncologie Medicale, Metz
  - CHRA;Hematologie, Metz-Tessy
  - Clinique Clementville; Hopital De Jour, Montpellier
  - Centre Azureen De Cancerologie; Cons externes, Mougins
  - Centre Antoine Lacassagne; B3 Medecine Conventionnelle, Nice
  - Hopital Cochin; Unite Fonctionnelle D Oncologie, Paris
  - Hopital Hotel Dieu; Oncologie Medicale, Paris
  - HOPITAL TENON; Cancerologie Medicale, Paris
  - Ch Francois Mitterrand; Medecine Oncologie, Pau
  - Ch Lyon Sud; Onco Secteur Jules Courmont, Pierre-Bénite
  - Chp Saint Gregoire; Cancerologie Radiotherapie, Saint-Grégoire
  - Ico Rene Gauducheau; Oncologie, Saint-Herblain
  - Clinique de L'Union; Oncologie, Saint-Jean
  - CMCO De La Cote D Opale; Auberge De Jour, Saint-Martin-Boulogne
  - Institut de Cancerologie de La Loire; Pneumologie, Saint-Priest-en-Jarez
  - Ch De Saint Quentin; Medecine B10, Saint-Quentin
  - Centre Paul Strauss; Oncologie Medicale, Strasbourg
  - Hopitaux Du Leman Site Thonon; Maternite Gynecologie, Thonon-les-Bains
  - Institut Claudius Regaud; Departement Oncologie Medicale, Toulouse
  - Clinique Pasteur; Pneumologie, Toulouse
  - Clinique Radio Des Dentellieres; Chimiotherapie Radiotherapie, Valenciennes
  - Centre-Alexis Vautrin, Vandœuvre-lès-Nancy
- Germany (54):
  - Klinikum Augsburg; Frauenklinik, Augsburg
  - Internist; Praxis Für Haemotologie & Onkologie, Bad Soden
  - Praxis Dres. Schilling & Till, Berlin
  - Vivantes Klinikum Am Urban; Zentrum für Brusterkrankungen, Berlin
  - Katholische Hospitalvereinigung Ostwestfalen gGmbH, Bielefeld
  - Gemeinschaftspraxis Dr. Bueckner und Dr. Nueckel, Bochum
  - Praxis Dr.med. Katja Ziegler-Löhr, Cologne
  - St. Elisabeth Krankenhaus Köln GmbH; Gynäkologie und Geburtshilfe, Cologne
  - Kliniken der Stadt Köln gGmbH Krankenhaus Holweide; Brustzentrum, Cologne
  - DONAU ISAR Klinikum Deggendorf; Frauenklinik, Deggendorf
  - Universitätsklinikum Essen; Zentrum Für Frauenheilkunde, Essen
  - Klinikum Essen-Mitte Ev. Huyssens-Stiftung / Knappschafts GmbH; Klinik für Senologie / Brustzentrum, Essen
  - Universitätsklinikum Freiburg; Frauenklinik, Freiburg im Breisgau
  - Klinikum St. Georg GmbH; Franziskus-Hospital Harderberg; Klinik für Gynaekologie und Geburtshilfe, Georgsmarienhütte
  - Krankenhaus St. Elisabeth und St. Barbara, Klinik für Frauenheilkunde und Geburtshilfe, Halle
  - Universitätsklinikum Hamburg-Eppendorf; Zentrum für operative Medizin Klinik für Gynäkologie, Hamburg
  - Kooperatives Mammazentrum Hamburg Krankenhaus Jerusalem, Hamburg
  - Gynaekologisch-Onkologische Schwerpunktpraxis Prof. Dr. med. Lueck, Dr. Schrader und Dr. Noeding, Hanover
  - Medizinische Hochschule Hannover, Klinik für Frauenheilkunde und Geburtshilfe, Hanover
  - Nationales Centrum für Tumorerkrankungen (NCT) ; Gyn. Onk. Frauenklinik; Uniklinikum Heidelberg, Heidelberg
  - Universitätsklinikum Jena; Klinik und Poliklinik für Frauenheilkunde und Fortpflanzungsmedizin, Jena
  - Elisabeth-Krankenhaus Brustzentrum, Kassel
  - Klinikum Kulmbach; Frauenklinik, Kulmbach
  - Dres. Andreas Köhler und Roswitha Fuchs, Langen
  - Klinikum Leverkusen; Med. Klinik III / Onkologie, Leverkusen
  - Klinikum Ludwigsburg; Klinik für Frauenheilkunde und Geburtshilfe, Ludwigsburg
  - Universitätsklinikum Schleswig-Holstein / Campus Lübeck; Klinik für Frauenheilkunde und Geburtshilfe, Lübeck
  - Onkologische Schwerpunktpraxis Lübeck, Lübeck
  - Universitätsmedizin Mainz; Klinik u. Poliklinik f. Geburtshilfe u. Frauenheilkunde, Mainz
  - Gemeinschaftspraxis Fr. Dr. med. Balser & Hr. Dr. med. Weidenbach, Marburg
  - Klinikum Meiningen Klinik f.Gynäkologie und Geburtshilfe, Meiningen
  - Klinikum Memmingen; Abt.Gynäkologie, Memmingen
  - Mühlenkreiskliniken; Johannes Wesling Klinikum Minden; Klinik für Frauenheilkunde und Geburtshilfe, Minden
  - Praxis Dr.med. Steffi Busch, Mühlhausen
  - Gemeinschaftspraxis Prof. Dr.med. Christoph Salat und Dr.med. Oliver J. Stötzer, München
  - Praxis Dr. Prechtl & Dr. Kowolik; Frauenklinik, München
  - Universitätsklinikum Münster; Klinik für Frauenheilkunde und Geburtshilfe, Münster
  - Ruppiner Kliniken, Klinik fuer Gynaekologie und Geburtshilfe, Neuruppin
  - Klinikum Nord Frauenklinik, Nuremberg
  - Sana Klinikum Offenbach GmbH; Klinik für Gynäkologie & Geburtshilfe, Offenbach
  - medius KLINIK OSTFILDERN-RUIT; Brustzentrum, Ostfildern
  - Oncologianova GmbH, Recklinghausen
  - Agaplesion Diakonieklinikum Rotenburg, Rotenburg (Wümme)
  - Caritas Klinik St. Theresia -Frauenklinik Brustzentrum, Saarbrücken
  - Leopoldina Krankenhaus der Stadt Schweinfurt GmbH, Schweinfurt
  - HELIOS Klinikum Schwerin; Frauenklinik, Schwerin
  - Johanniter-Krankenhaus Genthin-Stendal; Klinik Für Frauenheilkunde & Geburtshilfe, Stendal
  - Kreiskrankenhaus Torgau; Abt.Gynäkologie und Geburtshilfe, Torgau
  - Universitätsklinik Tübingen; Frauenklinik, Tübingen
  - Katharinen-Hospital gGmbH, Unna
  - GRN-Klinik Weinheim; Abt.Gynäkologie und Geburtshilfe, Weinheim
  - ASKLEPIOS KREISKRANKENHÄUSER WEIßENFELS-HOHENMÖLSEN GMBH, Weißenfels
  - Lahn-Dill Kliniken GmbH Klinikum Wetzlar Gynäkologie/Geburtshilfe, Wetzlar
  - Gesellschaft für Medizinische Studien Würselen, Würselen
- Greece (9):
  - Uni Hospital of Alexandroupoli; Dept. of Oncology - Duth, Alexandroupoli
  - Anticancer Hospital Ag Savas; 1St Dept of Internal Medicine, Athens
  - Laiko General Hospital; 1St Pathological Clinic, Athens
  - Alexandras General Hospital of Athens; Oncology Department, Athens
  - Periph. University General Hospital of Heraklion Crete; Oncology Department, Heraklion
  - Agioi Anargyroi Cancer Hospital; 2Nd Oncology Dept., Kifissia
  - University Hospital of Larissa; Oncology, Larissa
  - Euromedical General Clinic of Thessaloniki; Oncology Department, Thessaloniki
  - Papageorgiou General Hospital; Medical Oncology, Thessaloniki
- Guatemala (2):
  - Centro Oncológico Sixtino / Centro Oncológico SA, Guatemala City
  - Grupo Angeles, Guatemala City
- Hong Kong (2):
  - Queen Elizabeth Hospital; Clinical Oncology, Hong Kong
  - Prince of Wales Hosp; Dept. Of Clinical Onc, Shatin
- Hungary (8):
  - Szent Margit Hospital; Dept. of Oncology, Budapest
  - Szent Imre Hospital; Dept. of Oncology, Budapest
  - Orszagos Onkologiai Intezet, Budapest
  - Semmelweis Egyetem Aok; Iii.Sz. Belgyogyaszati Klinika, Budapest
  - Debreceni Egyetem Klinikai Kozpont ; Department of Oncology, Debrecen
  - Josa Andras Korhaz; Dept of Oncoradiology, Nyíregyháza
  - Pécsi Tudományegyetem; Klinikai Központ Onkoterápiás Intézet, Pécs
  - Markusovszky Hospital, Szombathely
- Indonesia (5):
  - Hasan Sadikin Hospital; Internal Medicine, Bandung
  - CiptoMangunkusumo Hospital; Internal Medicine, Central Jakarta
  - Soetomo Hospital; Surgery, East Java
  - Dharmais National Cancer Center, Jakarta
  - Sardjito Hospital; Instalasi Kanker Tulip, Yogyakarta
- Ireland (6):
  - Mater Misericordiae Uni Hospital; Oncology, Dublin
  - Mater Private Hospital, Dublin
  - Beaumont Hospital; Cancer Clinical Trials Unit, Dublin
  - University Hospital Limerick, Limerick
  - Sligo General Hospital; Oncology, Sligo
  - Waterford Regional Hospital; Department Of Medical Oncology, Waterford
- Italy (31):
  - Irccs Ist. Tumori Giovanni Paolo Ii; Dipartimento Oncologia Medica, Bari, Apulia
  - Ospedale Vito Fazzi; Div. Oncoematologia, Lecce, Apulia
  - IRCCS Ospedale Casa Sollievo Della Sofferenza; Oncologia, San Giovanni Rotondo, Apulia
  - Ospedale Oncologico Regionale; U.O. Oncologia Medica Ed Ematologia, Rionero in Vulture, Basilicate
  - Azienda Ospedaliera A. Cardarelli, Napoli, Campania
  - Istituto Nazionale Tumori Irccs Fondazione g. PASCALE;U.O.C. Oncologia Medica Senologica, Napoli, Campania
  - Università degli Studi Federico II; Clinica di Oncologia Medica, Napoli, Campania
  - IRST Istituto Scientifico Romagnolo Per Lo Studio E Cura Dei Tumori, Sede Meldola; Oncologia Medica, Meldola, Emilia-Romagna
  - Ospedale Regionale Di Parma; Divisione Di Oncologia Medica, Parma, Emilia-Romagna
  - Az. Osp. Ospedale Civile; U.O. Di Oncologia Medica Ed Ematologia, Piacenza, Emilia-Romagna
  - Azienda USL di Ravenna; Unità Operativa di Oncologia Medica, Ravenna, Emilia-Romagna
  - Ausl Frosinone - Ospedale Umberto I; Divisione Di Oncologia, Frosinone, Lazio
  - IFO - Istituto Regina Elena; Oncologia Medica, Rome, Lazio
  - Policlinico Umberto i di Roma; dip. Scienze Radiologiche, Oncologiche, Anatomopatologiche, Rome, Lazio
  - Azienda Ospedaliera Sant'Andrea, Rome, Lazio
  - Ospedale Belcolle Di Viterbo; Oncologia, Viterbo, Lazio
  - Asst Papa Giovanni XXIII; Oncologia Medica, Bergamo, Lombardy
  - ASST DI CREMONA; Unità di Patologia Mammaria Senologia e Breast Unit, Cremona, Lombardy
  - Fondazione IRCCS Istituto Nazionale dei Tumori; S. C. Oncologia Medica 2, Milan, Lombardy
  - ASST DI MONZA; Oncologia Medica, Monza, Lombardy
  - IRRCCS San Matteo; Dip Oncoematologico ; Divisione Oncologia, Pavia, Lombardy
  - IRCCS Istituto Clinico Humanitas; Oncologia, Rozzano, Lombardy
  - A.O. Città della Salute e della Scienza - Presidio Molinette; divisione oncologia medica, Turin, Piedmont
  - Ospedale Oncologico A.Businco; Div. Oncologia Medica II, Cagliari, Sardinia
  - Ospedale Civile SS Annunziata; oncologia medica, Sassari, Sardinia
  - Ospedale Garibaldi Nesima; Biomedicina Clinica e Molecolare, Catania, Sicily
  - Azienda Ospedaliero-Universitaria Careggi;S.C. Oncologia Medica 1, Florence, Tuscany
  - Azlenda Ospendaliero-Universitaria Pisana; C.O. Oncologia 2, Pisa, Tuscany
  - Azienda usl 5 Di Pisa-Ospedale Di Pontedera;U.O. Oncologia, Pontedera, Tuscany
  - Ospedale Civile; Oncologia Medica, Camposampiero, Veneto
  - Arcispedale S.Anna; Oncologia Medica, Cona (Ferrara), Veneto
- Lithuania (2):
  - Hospital of Lithuanian University of Health. Sciences Kaunas Clinics, Kaunas
  - Klaipeda University Hospital, Klaipėda
- Malaysia (4):
  - Hospital Wanita dan Kanak-Kanak Sabah, Sabah, Sabah
  - Sarawak General Hospital; Department of Radiotherapy, Oncology and Palliative care, Sarawak, Sarawak
  - Hospital Pulau Pinang; Jabatan Radioterapi & Onkologi, George Town
  - University Malaya Medical Centre; Clinical Oncology Unit,, Kuala Lumpur
- Mexico (7):
  - Centro Estatal de Oncología de Campeche, Campeche
  - Centro Estatal de Cancerología, Chihuahua City
  - Instituto Nacional de Cancerologia; Oncology, Distrito Federal
  - Consultorio de Medicina Especializada; Dentro de Condominio San Francisco, Mexico City
  - Oaxaca Site Management Organization, Oaxaca City
  - Cancerologia de Queretaro; Oncologia, Queretaro, Queretaro
  - Centro Estatal de Cancerologia de Nayarit, Tepic
- Institut National D'oncologie Sidi Med Benabdellah, Rabat, Morocco
- Netherlands (20):
  - Jeroen Bosch Ziekenhuis, 's-Hertogenbosch
  - Onze Lieve Vrouwe Gasthuis, AC Amsterdam
  - Gelre Ziekenhuis Apeldoorn, Lokatie Lukas; Afdeling Interne Geneeskunde, Apeldoorn
  - Rijnstate Ziekenhuis; Inwendige Geneeskunde, Arnhem
  - Albert Schweitzer Ziekenhuis - loc Dordrecht, Dordrecht
  - Ziekenhuis Gelderse Vallei; Inwendige Geneeskunde, Ede
  - Catharina Ziekenhuis; Dept of Internal Medicin, Eindhoven
  - Maxima Medisch Centrum; Inwendige Geneeskunde, Eindhoven
  - Martini Ziekenhuis; Dept of Internal Medicine, Groningen
  - Atrium Medisch Centrum Parkstad, Heerlen, Heerlen
  - Spaarne Ziekenhuis; Inwendige Geneeskunde, Hoofddorp
  - St. Antonius Ziekenhuis Nieuwegein, Nieuwegein
  - Franciscus Ziekenhuis, Roosendaal
  - Maasstad ziekenhuis; Afdeling oncologie hematologie, Rotterdam
  - Ikazia Ziekenhuis, Rotterdam
  - Vlietland Ziekenhuis, Locatie Schiedam; Interne Geneeskunde, Schiedam
  - Zuyderland ziekenhuis locatie Geleen, Sittard-Geleen
  - Diakonessenhuis Utrecht: ziekenhuisapotheek, Utrecht
  - Ziekenhuis VieCurie Vitaal, Venlo
  - Zaans Medisch Centrum, Zaandam
- Tauranga Hospital, Clinical Trials Unit; BOP Clinical School, Tauranga, New Zealand
- Norway (3):
  - Sørlandet Sykehus Kristiansand, Kristiansand
  - Oslo universitetssykehus HF, Ullevål, Kreftsenteret, Oslo
  - Helse Stavanger HF, Stavanger Universitetssjukehus; Klinikk for Blod og kreftsykdommer, Stavanger
- Pakistan (4):
  - Shifa International Hospital; Department of Oncology, Islamabad
  - Aga Khan University; Department of Oncology, Karachi
  - Shaukat Khanum Memorial Cancer Hospital; Department of Oncology, Lahore
  - Hameed Latif Hospital; Department of Oncology, Lahore
- Centro Hemato Oncologico Panama, Panama City, Panama
- Peru (5):
  - Centro Medico Monte Carmelo, Arequipa
  - Instituto Nacional de Enfermedades Neoplasicas, Lima
  - Clinica de Especialidades Medicas, Lima
  - Clinica Internacional, Sede San Borja; Unidad de Investigacion de Clínica Internacional, Lima
  - Instituto Oncologico de Lima, Lima
- Philippines (2):
  - Philippine General Hospital; Section Of Medical Oncology, Manila
  - East Avenue Medical Center, Quezon City
- Poland (7):
  - Poradnia Onkologiczna oraz Oddzial Kliniczny Onkologii SPZOZ Szpital Uniwersytecki, Krakow
  - Europejskie Centrum Zdrowia Otwock Szpital im. Fryderyka Chopina, Klinika Onkologii, Otwock
  - Oddzial Chemioterapii Szpitala Klinicznego Nr 1 w Poznaniu, Poznan
  - Wielkopolskie Centrum Onkologi, Poznan
  - MRUKMED Lekarz Beata Madej-Mruk i Partner Spolka Partnerska Oddzial nr 1 w Rzeszowie, Rzeszów
  - Wojewodzki Szpital Zespolony, Torun
  - NZOZ Onko-Dent SP. P. G. L. Slomian, Poradnia Onkologiczna, Żory
- Portugal (4):
  - Centro Clinico Champalimaud; Oncologia Medica, Lisbon
  - Hospital da Luz; Departamento de Oncologia Medica, Lisbon
  - IPO do Porto; Servico de Oncologia Medica, Porto
  - Hospital de Sao Joao; Servico de Oncologia, Porto
- Romania (9):
  - Policlinica Sfanta Maria - Oncology; Medical Oncology, Baia Mare
  - Institut of Oncology Al. Trestioreanu Bucharest; Oncology Department, Bucharest
  - Emergency University Bucharest Hospital; Oncology Department, Bucharest
  - Cluj Clinical County Hospital; Oncology Dept, Cluj-Napoca
  - Prof. Dr. I. Chiricuta Institute of Oncology, Cluj-Napoca
  - SC Oncolab SRL, Craiova
  - Clinical Hospital 1 Craiova; Medical Oncology, Craiova
  - S.C. Life Search S.R.L; Medical Oncology Clinic, Timișoara
  - ONCOMED - Medical Centre, Timișoara
- Russia (7):
  - Regional Oncology Hospital, Irkutsk
  - City Oncological Hospital, Izhevsk
  - Russian Oncology Research Center n.a. N.N. Blokhin Dpt of Clinical Pharmacology and Chemotherapy, Moscow
  - City Clinical Oncology Hospital, Moscow
  - State Inst. Of Healthcare Orenburg Regional Clinical Oncology Dis, Orenburg
  - City Clinical Oncology Dispensary, SPb SBIH CCOD, Saint Petersburg
  - Bashkirian Republican Clinical Oncology Dispensary, Ufa
- Saudi Arabia (2):
  - King Faisal Specialist Hospital & Research Centre, Jeddah
  - King Abdul Aziz Medical City, King Fahd National Guard; Oncology, Riyadh
- Serbia (5):
  - Clinical Hospital Center Bezanijska kosa; Clinic for Oncology, Belgrade
  - Institute for Onc/Rad Serbia, Belgrade
  - Oncology Institute of Vojvodina, Kamenitz
  - Clinical Center Kragujevac, Kragujevac
  - Clinical Centre Nis, Clinic for Oncology, Niš
- National Cancer Centre; Medical Oncology, Singapore, Singapore
- Slovakia (5):
  - Mammacentrum sv. Agáty, Banská Bystrica
  - National Cancer Institute - Comenius University; Dept. Clinical Oncology, Bratislava
  - Vychodoslovensky onkologicky ustav, Košice
  - Fakultna nemocnica s poliklinikou J.A. Reimana Presov, Prešov
  - Fakultna nemocnica Trencín; Onkologicke odd., Trenčín
- University Medical Centre Maribor; Depart. of Gynecology & Breast Oncology, Maribor, Slovenia
- South Africa (3):
  - Westridge Medical Center, Durban
  - Donald Gordon Medical Centre, Johannesburg
  - Steve Biko Academic Hospital; Oncology, Pretoria
- South Korea (5):
  - National Cancer Center, Goyang-si
  - Samsung Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Yonsei University Severance Hospital; Medical Oncology, Seoul
  - Asan Medical Center., Seoul
- Spain (33):
  - Hospital General de Elda; Servicio de Oncologia, Elda, Alicante
  - Hospital Universitario Son Espases, Palma de Mallorca, Balearic Islands
  - Hospital Universitari Germans Trias i Pujol; Servicio de Oncologia, Badalona, Barcelona
  - Corporacio Sanitaria Parc Tauli; Servicio de Oncologia, Sabadell, Barcelona
  - Hospital Universitario Marques de Valdecilla; Servicio de Oncologia, Santander, Cantabria
  - IInstituto Oncologico de San Sebastian, Oncologikoa; Servicio de Oncologia, Donostia / San Sebastian, Guipuzcoa
  - Hospital Universitario Materno Infantil de Gran Canaria; Servicio de Oncologia, Las Palmas de Gran Canaria, LAS Palmas
  - Hospital de Gran Canaria Dr. Negrin; Servicio de Oncologia, Las Palmas de Gran Canaria, LAS Palmas
  - Hospital Quiron de Madrid; Servicio de Oncologia, Pozuelo de Alarcón, Madrid
  - Hospital de Navarra; Servicio de Oncologia, Navarra, Navarre
  - Hospital Do Meixoeiro; Servicio de Oncologia, Vigo, Pontevedra
  - Hospital de Cabueñes; Servicio de Oncologia, Gijón, Principality of Asturias
  - Hospital Universitario de Canarias;servicio de Oncologia, San Cristóbal de La Laguna, Tenerife
  - Complejo Hospitalario Nuestra Señora de la Candelaria; Servicio de Oncologia, Santa Cruz de Tenerife, Tenerife
  - Hospital Lluis Alcanys; Servicio de Oncologia, Xàtiva, Valencia
  - Hospital de Basurto; Servicio de Oncologia, Bilbao, Vizcaya
  - Complejo Hospitalario Universitario de Albacete; Servicio de Oncologia, Albacete
  - Hospital General Univ. de Alicante; Servicio de Oncologia, Alicante
  - Hospital del Mar; Servicio de Oncologia, Barcelona
  - Hospital de la Santa Creu i Sant Pau; Servicio de Oncologia, Barcelona
  - Hospital Duran i Reynals; Oncologia, Barcelona
  - Complejo Asistencial Universitario De Burgos; Servicio de Oncologia, Burgos
  - Hospital San Pedro De Alcantara; Servicio de Oncologia, Cáceres
  - Complejo Hospitalario de Jaen-Hospital Universitario Medico Quirurgico; Servicio de Oncologia, Jaén
  - Complejo Asistencial Universitario de Leon; Servicio de Oncologia, León
  - Hospital Universitari Arnau de Vilanova de Lleida; Servicio de Oncologia, Lleida
  - Hospital Ramon y Cajal; Servicio de Oncologia, Madrid
  - Hospital Universitario Clínico San Carlos; Servicio de Oncologia, Madrid
  - HOSPITAL DE MADRID NORTE SANCHINARRO- CENTRO INTEGRAL ONCOLOGICO CLARA CAMPAL; Servicio de Oncologia, Madrid
  - Hospital Universitario Virgen de Arrixaca; Servicio de Oncologia, Murcia
  - Complejo Hospitalario de Toledo- H. Virgen de la Salud; Servicio de Oncologia, Toledo
  - Hospital Arnau de Vilanova (Valencia) Servicio de Oncologia, Valencia
  - Hospital Clinico Universitario Lozano Blesa; Servicio de Oncologia, Zaragoza
- Sweden (2):
  - Skånes University Hospital, Skånes Department of Onclology, Lund
  - Skaraborgs sjukhus Skoevde, Dept of surgery, Skövde
- Switzerland (9):
  - Hirslanden Medical Center, Tumorzentrum, Aarau
  - Kantonsspital Baden; Frauenklinik, Baden
  - Ospedale San Giovanni; Oncologia, Bellinzona
  - Inselspital Bern; Universitätsklinik für medizinische Onkologie, Bern
  - Kantonsspital Frauenfeld, Frauenklinik Thurgau, Frauenfeld
  - CHUV; Departement d'Oncologie, Lausanne
  - Spital Thun; Medizinische Klinik, Thun
  - Kantonsspital Winterthur; Medizinische Onkologie, Winterthur
  - Stadtspital Triemli; Frauenklinik, Zurich
- Taiwan (4):
  - China Medical University Hospital; Surgery, Taichung
  - National Cheng Kung Uni Hospital; Surgery, Tainan
  - National Taiwan Uni Hospital; General Surgery, Taipei
  - Tri-Service General Hospital, Division of General Surgery, Taipei
- Thailand (6):
  - Department of Surgery, King Chulalongkorn Memorial Hospital, Bangkok
  - Pramongkutklao Hospital; Medicine - Medical Oncology Unit, Bangkok
  - Rajvithi Hospital, Bangkok
  - Ramathibodi Hospital; Medicine/Oncology, Bangkok
  - Maharaj Nakorn Chiang Mai Hospital; Department of Surgery/Head Neck and Breast Unit; Clinical Trial, Chiang Mai
  - Oncology Unit, Faculty of Medicine, Vajira Hospital; Department of Medicine, Dusit
- Turkey (Türkiye) (10):
  - Ankara Uni School of Medicine; Medical Oncology, Ankara
  - Akdeniz University Medical Faculty; Medical Oncology Department, Antalya
  - Dicle University Faculty of Medicine, Diyarbakır
  - Gaziantep Univ. Med. Fac., Gaziantep
  - Istanbul Uni of Medicine Faculty; Oncology Dept, Istanbul
  - Marmara Uni Faculty of Medicine; Medical Oncology, Istanbul
  - Kocaeli University Faculty of Medicine; Medical oncology, İzmit
  - Mersin University Medical Faculty, Mersin
  - 19 Mayis University Medical Faculty; Medical Oncology Department, Samsun
  - Hacettepe Uni Medical Faculty Hospital; Oncology Dept, Sihhiye/Ankara
- Ukraine (2):
  - Kyiv City Clinical Oncological Center; Chemotherapy Department, Kiev
  - State Oncology Regional Treatment-Diagnostic Center; Chemotherapy Department, Lviv
- Tawam Hospital, Al Ain City, United Arab Emirates
- United Kingdom (50):
  - Nevill Hall Hospital, Abergavenny
  - Bedford Hospital; Oncology, Bedford
  - Wexham Park Hospital; Oncology, Berkshire
  - University Hospital Birmingham Queen Elizabeth Hospital, Birmingham
  - Heartlands Hospital; Department Of Medicine, Birmingham
  - Royal Bournemouth Hospital; Oncology, Bournemouth
  - Kent & Canterbury Hospital, Canterbury
  - Broomfield Hospital; Oncology, Chelmsford
  - Glan Clwyd Distr Gen Hospital;Nth Wales Cancer Treatment Ctr, Denbighshire
  - Royal Derby Hospital, Derby
  - North Devon District Hospital, Devon
  - Russells Hall Hospital; Oncology, Dudley
  - University Hospital of North Durham, Durham
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Inverclyde Hospital, Greenock
  - Diana Princess of Wales Hosp., Grimsby
  - Royal Surrey County Hospital, Guildford
  - Princess Alexandra Hospital; Oncology Department, Harlow
  - Huddersfield Royal Infirmary, Huddersfield
  - Ipswich Hospital, Ipswich
  - Crosshouse Hospital; Dept of Oncology, Kilmarnock
  - Forth Valley Royal Hospital ; Oncology Department, Larbert
  - Leicester Royal Infirmary, Leicester
  - St John's Hospital, Livingston
  - Guys and St Thomas NHS Foundation Trust, Guys Hospital, London
  - Queen Elizabeth Hospital, London
  - St George's Hospital, London
  - Macclesfield District General Hospital, Macclesfield
  - Christie Hospital; Breast Cancer Research Office, Manchester
  - The Clatterbridge Cancer Ctr For Oncolgy, Metropolitan Borough of Wirral
  - Freeman Hospital; Northern Centre For Cancer Care, New Castle Upon Tyne
  - Royal Gwent Hospital, Newport
  - North Tyneside General Hospital, North Shields
  - Northampton General Hospital NHS Trust, Northampton
  - Derriford Hospital; Plymouth Oncology Centre, Plymouth
  - Poole General Hospital, Poole
  - Queen Alexandra Hospital, Portsmouth, Portsmouth
  - Royal Preston Hospital, Preston
  - Queens Hospital; R&D, Romford
  - Scarborough General Hospital, Scarborough
  - Royal Shrewsbury Hospital; Pharmacy Department, Shrewsbury
  - Southampton General Hospital, Southampton
  - Sunderland Royal Hospital, Sunderland
  - Singleton Hospital; Pharmacy Department, Swansea
  - Great Western Hospital, Swindon Cancer Research Unit; Osprey Unit Level 3, Swindon
  - Royal Cornwall Hospital, Truro
  - Royal Hampshire County Hospital; Winchester & Andover Breast Unit, Winchester
  - The Royal Wolverhampton Hospitals NHS Trust, Wolverhampton
  - Airedale General Hospital; Oncology, York
  - York District Hospital, York
- Uruguay (3):
  - Grupo Oncológico Cooperativo Uruguayo; Hospital de Clínicas - Dpto. de Oncología, Montevideo
  - Hospital Militar; Oncologia, Montevideo
  - Hospital Pereira Rossell; Oncology Department, Montevideo
- Venezuela (3):
  - Instituto Oncológico Luis Razetti, Caracas
  - Centro Integral de Oncología, Caracas
  - Centro Médico Docente La Trinidad; Unidad de Protocolos Clínicos, Caracas
- K hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.clinicalstudydatarequest.com). Further details on Roche's criteria for eligible studies are available here (https://clinicalstudydatarequest.com/Study Sponsors/Study-Sponsors-Roche.aspx). For further details on Roche's Global Policy on Sharing of Clinical Study Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Jung KH, Ataseven B, Verrill M, Pivot X, De Laurentiis M, Al-Sakaff N, Lauer S, Shing M, Gligorov J, Azim HA. Adjuvant Subcutaneous Trastuzumab for HER2-Positive Early Breast Cancer: Subgroup Analyses of Safety and Active Medical Conditions by Body Weight in the SafeHer Phase III Study. Oncologist. 2018 Oct;23(10):1137-1143. doi: 10.1634/theoncologist.2018-0065. Epub 2018 Jul 17. PMID 30018134
- [Derived] Gligorov J, Ataseven B, Verrill M, De Laurentiis M, Jung KH, Azim HA, Al-Sakaff N, Lauer S, Shing M, Pivot X; SafeHer Study Group. Safety and tolerability of subcutaneous trastuzumab for the adjuvant treatment of human epidermal growth factor receptor 2-positive early breast cancer: SafeHer phase III study's primary analysis of 2573 patients. Eur J Cancer. 2017 Sep;82:237-246. doi: 10.1016/j.ejca.2017.05.010. Epub 2017 Jun 16. PMID 28625777

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 2984 participants screened, a total of 2577 participants were enrolled into the trial, and 2573 participants received at least one dose of study treatment.
  4 Participants were not included in the Safety Follow-Up (SFU) ITT due to the lack of Principal Investigator signatures.
Groups:
- Cohort A: SC Herceptin by Needle/Syringe: Participants received SC Herceptin by an assisted administration as 600 mg every 3 weeks for a total of 18 doses/cycles. Each dose of SC Herceptin was taken from a single-use vial and injected by needle/syringe.
- Cohort B: SC Herceptin by Single-Use Injection Device (SID): Participants received SC Herceptin as 600 mg every 3 weeks for a total of 18 doses/cycles. Each dose of SC Herceptin was administered from a pre-filled SID. The first administration was performed by a healthcare professional (HCP). Subsequent doses were self-administered by participants who were willing and judged competent by the HCP.
Period: Treatment Period
Arm/Group | Cohort A: SC Herceptin by Needle/Syringe | Cohort B: SC Herceptin by Single-Use Injection Device (SID)
Started | 1867 | 710
Completed | 1670 | 652
Not Completed | 197 | 58
Not completed — Withdrawal by Subject | 35 | 9
Not completed — Disease Progression/Recurrence | 37 | 13
Not completed — Investigator/Sponsor Decision | 6 | 3
Not completed — Other | 13 | 2
Not completed — Lack of Compliance | 5 | 1
Not completed — Adverse Event | 100 | 30
Not completed — Pregnancy | 1 | 0
Period: Safety Follow-up
Arm/Group | Cohort A: SC Herceptin by Needle/Syringe | Cohort B: SC Herceptin by Single-Use Injection Device (SID)
Started | 1865 (Participants who discontinued treatment were allowed to join the SFU Period.) | 708 (Participants who discontinued treatment were allowed to join the SFU Period.)
Completed | 1318 | 501
Not Completed | 547 | 207
Not completed — Physician Decision | 6 | 4
Not completed — Lost to Follow-up | 101 | 48
Not completed — Withdrawal by Subject | 155 | 49
Not completed — Death | 28 | 4
Not completed — Non-compliance | 7 | 3
Not completed — Protocol Violation | 7 | 0
Not completed — Site closure | 2 | 3
Not completed — Erroneous reporting or late reporting | 2 | 0
Not completed — Missing | 7 | 2
Not completed — Disease progression /disease recurrence | 223 | 90
Not completed — Sponsor decision | 1 | 0
Not completed — Adverse Event | 8 | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: All participants enrolled into the study regardless of whether treatment was received.
Groups:
- Cohort B: SC Herceptin by SID: Participants received SC Herceptin as 600 mg every 3 weeks for a total of 18 doses/cycles. Each dose of SC Herceptin was administered from a pre-filled SID. The first administration was performed by an HCP. Subsequent doses were self-administered by participants who were willing and judged competent by the HCP.
- Total: Total of all reporting groups
Arm/Group | Cohort A: SC Herceptin by Needle/Syringe | Cohort B: SC Herceptin by SID | Total
Number analyzed (Participants) | 1867 | 710 | 2577
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (12.01) | 53.0 (11.32) | 53.7 (11.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1863 | 710 | 2573
  Male | 4 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With At Least 1 Adverse Event (AE) During the Treatment Period
Description: Participants were planned to receive a total of 18 cycles of SC Herceptin. An AE was defined as any untoward medical occurrence in a participant administered SC Herceptin. Examples included unfavorable/unintended signs and symptoms, new or exacerbated disease, recurrence of intermittent condition, deterioration in laboratory value or other clinical test, or adverse procedure-related events. The percentage of participants with at least 1 AE during the treatment period (regardless of severity or seriousness) was reported.
Time Frame: From Day 1 up to 19 cycles (cycle length 3 weeks) (approximately 1 year)
Population: Safety Population: All enrolled participants who received at least one dose of study medication according to assigned treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: SC Herceptin by Needle/Syringe | Cohort B: SC Herceptin by SID
Number analyzed (Participants) | 1864 | 709
percentage of participants | 88.6 | 89.0

2. Primary Outcome: Percentage of Participants With a Grade 3 or Higher AE During the Treatment Period
Description: Participants were planned to receive a total of 18 cycles of SC Herceptin. An AE was defined as any untoward medical occurrence in a participant administered SC Herceptin. Examples included unfavorable/unintended signs and symptoms, new or exacerbated disease, recurrence of intermittent condition, deterioration in laboratory value or other clinical test, or adverse procedure-related events. AEs were graded according to National Cancer Institute Common Terminology Criteria Version 4.0. Grade 3 AEs were those considered severe or medically significant but not immediately life-threatening. Grade 4 AEs were those considered life-threatening and/or for which urgent intervention was indicated. Grade 5 AEs were those resulting in death. The percentage of participants with a Grade 3 or higher (i.e., Grade 3 to 5) AE during the treatment period was reported.
Time Frame: From Day 1 up to 19 cycles (cycle length 3 weeks) (approximately 1 year)
Population: Safety Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: SC Herceptin by Needle/Syringe | Cohort B: SC Herceptin by SID
Number analyzed (Participants) | 1864 | 709
percentage of participants | 24.0 [22.1 to 26.0] | 21.0 [18.1 to 24.2]

3. Primary Outcome: Percentage of Participants With Treatment Interruption Due to an AE
Description: Participants were planned to receive a total of 18 cycles of SC Herceptin. An AE was defined as any untoward medical occurrence in a participant administered SC Herceptin. Examples included unfavorable/unintended signs and symptoms, new or exacerbated disease, recurrence of intermittent condition, deterioration in laboratory value or other clinical test, or adverse procedure-related events. The percentage of participants with SC Herceptin treatment interrupted to assess or treat AEs was reported.
Time Frame: From Day 1 up to 19 cycles (cycle length 3 weeks) (approximately 1 year)
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: SC Herceptin by Needle/Syringe | Cohort B: SC Herceptin by SID
Number analyzed (Participants) | 1864 | 709
percentage of participants | 9.8 | 10.4

4. Primary Outcome: Number of Herceptin Cycles Received
Description: Participants were planned to receive a total of 18 cycles of SC Herceptin. The median number of cycles actually received was reported.
Time Frame: From Day 1 up to 19 cycles (cycle length 3 weeks) (approximately 1 year)
Population: Safety Population. The endpoint also included an analysis of a subgroup of participants from Cohort B who received doses of self-administered SC Herceptin via SID.
Measure: Median (Full Range); unit: cycles
Groups:
- Cohort B: SC Herceptin by SID (Self-Administered): Participants received SC Herceptin as 600 mg every 3 weeks for a total of 18 doses/cycles. Each dose of SC Herceptin was administered from a pre-filled SID. Dosing was either performed by self-administration or a qualified HCP. The present subgroup included only participants for whom SC Herceptin was given by self-administration.
Arm/Group | Cohort B: SC Herceptin by SID (Self-Administered) | Cohort A: SC Herceptin by Needle/Syringe | Cohort B: SC Herceptin by SID
Number analyzed (Participants) | 550 | 1864 | 709
cycles | 16.0 [1 to 17] | 18.0 [1 to 19] | 18.0 [1 to 18]

5. Primary Outcome: Percentage of Participants by Total Number of Herceptin Cycles Received
Description: Participants were planned to receive a total of 18 cycles of SC Herceptin. The percentage of participants was reported by the total number of cycles actually received. Because the data are presented non-cumulatively, this table reflects participant distribution by the highest number of cycles received.
Time Frame: From Day 1 up to 19 cycles (cycle length 3 weeks) (approximately 1 year)
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Groups:
- Cohort B: SC Herceptin by SID (Self- Administered): Participants received SC Herceptin as 600 mg every 3 weeks for a total of 18 doses/cycles. Each dose of SC Herceptin was administered from a pre-filled SID. Dosing was either performed by self-administration or a qualified HCP. The present subgroup included only participants for whom SC Herceptin was given by self- administration.
Arm/Group | Cohort B: SC Herceptin by SID (Self- Administered) | Cohort A: SC Herceptin by Needle/Syringe | Cohort B: SC Herceptin by SID
Number analyzed (Participants) | 550 | 1864 | 709
percentage of participants
  1 Cycle Received | 2.7 | 1.0 | 0.8
  2 Cycles Received | 1.3 | 0.5 | 0.4
  3 Cycles Received | 1.1 | 0.5 | 0.1
  4 Cycles Received | 1.6 | 1.2 | 0.7
  5 Cycles Received | 1.3 | 0.8 | 0.6
  6 Cycles Received | 1.6 | 0.5 | 0.1
  7 Cycles Received | 2.2 | 0.7 | 0.8
  8 Cycles Received | 2.2 | 0.9 | 0.3
  9 Cycles Received | 1.8 | 0.2 | 0.6
  10 Cycles Received | 1.5 | 0.3 | 0.1
  11 Cycles Received | 3.5 | 0.4 | 0.3
  12 Cycles Received | 2.5 | 0.9 | 0.8
  13 Cycles Received | 4.9 | 0.2 | 0
  14 Cycles Received | 6.9 | 0.5 | 0.6
  15 Cycles Received | 10.7 | 0.5 | 0.4
  16 Cycles Received | 21.6 | 0.6 | 0.3
  17 Cycles Received | 32.5 | 1.0 | 1.1
  18 Cycles Received | 0 | 89.2 | 91.8
  19 Cycles Received | 0 | 0.2 | 0

6. Primary Outcome: Percentage of Participants Who Received Concomitant Cancer Therapy
Description: Concomitant cancer treatment included chemotherapy, radiotherapy, and hormone therapy administered during the study. The percentage of participants who received any of these concomitant therapies was reported.
Time Frame: From Baseline to data cutoff of 10 March 2015 (up to approximately 3 years)
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: SC Herceptin by Needle/Syringe | Cohort B: SC Herceptin by SID
Number analyzed (Participants) | 1864 | 709
percentage of participants
  Chemotherapy | 58.2 | 63.9
  Radiotherapy | 51.3 | 48.5
  Hormone Therapy | 53.5 | 50.4

7. Primary Outcome: Percentage of Participants Who Received Concomitant Non-Cancer Therapy
Description: Concomitant non-cancer treatment included any pharmacologic interventions administered during the study other than chemotherapy, radiotherapy, or hormone therapy. The percentage of participants who received any concomitant non-cancer therapies was reported.
Time Frame: From Baseline to data cutoff of 10 March 2015 (up to approximately 3 years)
Population: Safety Population
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: SC Herceptin by Needle/Syringe | Cohort B: SC Herceptin by SID
Number analyzed (Participants) | 1864 | 709
percentage of participants | 89.1 | 89.7

8. Secondary Outcome: Percentage of Participants Who Died by Data Cutoff of 10 March 2015
Description: The percentage of participants who died from any cause was reported.
Time Frame: From Baseline to time of event (maximum follow-up approximately 3 years as of data cutoff of 10 March 2015)
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Cohort A: SC Herceptin by Needle/Syringe | Cohort B: SC Herceptin by SID
Number analyzed (Participants) | 1867 | 710
percentage of participants | 1.5 | 0.8

9. Secondary Outcome: Percentage of Participants Who Died During the Safety Follow-up Period
Description: The percentage of participants who died from any cause was reported during the safety follow-up period.
Time Frame: From Baseline to Time of Event, Safety Follow-Up Period (Up to 6 Years)
Population: ITT Population
Measure: Number; unit: Percentage of Participants
Arm/Group | Cohort A: SC Herceptin by Needle/Syringe | Cohort B: SC Herceptin by SID
Number analyzed (Participants) | 1865 | 708
Percentage of Participants | 6.8 | 7.3

10. Secondary Outcome: Disease-Free Survival Rate
Description: DFS is defined as the time from first dose of SC Herceptin to the first event of local, regional or distant recurrence, contralateral invasive breast cancer (including ipsilateral ductal carcinoma in situ) or death due to any cause.
  Time from the date of first dose to any DFS event was expressed in Kaplan-Meier survival probability estimates. Patients without an event will be censored at the last assessment date.
Time Frame: From Baseline to time of event (up to approximately 8 years)
Population: ITT Population who completed Safety Follow-up
Measure: Number (95% Confidence Interval); unit: Kaplan-Meier survival probability
Arm/Group | Cohort A: SC Herceptin by Needle/Syringe | Cohort B: SC Herceptin by SID
Number analyzed (Participants) | 1865 | 708
Kaplan-Meier survival probability
  0.5 Year | 0.990 [0.984 to 0.993] | 0.987 [0.976 to 0.993]
  1 Year | 0.975 [0.967 to 0.981] | 0.976 [0.961 to 0.985]
  1.5 Year | 0.960 [0.950 to 0.968] | 0.957 [0.939 to 0.970]
  2 Years | 0.934 [0.921 to 0.944] | 0.939 [0.918 to 0.955]
  3 Years | 0.904 [0.889 to 0.917] | 0.896 [0.870 to 0.916]
  4 Years | 0.881 [0.865 to 0.896] | 0.874 [0.847 to 0.897]
  5 Years | 0.868 [0.851 to 0.883] | 0.863 [0.835 to 0.887]
  6 Years | 0.851 [0.833 to 0.867] | 0.853 [0.824 to 0.878]

11. Secondary Outcome: Overall Survival Rate
Description: Overall survival was defined as the time from randomization to death from any cause.
  Time from the date of randomization to the date of death was expressed in Kaplan-Meier survival probability estimates. Patients without an event will be censored at the last assessment date.
Time Frame: From Baseline to Time of Event (Up to Approximately 6 Years)
Population: ITT population: All randomized participants received at least one dose of drug and completed the follow up period
Measure: Number (95% Confidence Interval); unit: Kaplan-Meier survival probability
Groups:
- Cohort B: SC Herceptin by SIDE: Participants received SC Herceptin as 600 mg every 3 weeks for a total of 18 doses/cycles. Each dose of SC Herceptin was administered from a pre-filled SID. The first administration was performed by an HCP. Subsequent doses were self-administered by participants who were willing and judged competent by the HCP.
Arm/Group | Cohort A: SC Herceptin by Needle/Syringe | Cohort B: SC Herceptin by SIDE
Number analyzed (Participants) | 1865 | 708
Kaplan-Meier survival probability
  0.5 Year | 0.999 [0.996 to 1.000] | 0.996 [0.987 to 0.999]
  1 Year | 0.998 [0.994 to 0.999] | 0.994 [0.985 to 0.998]
  1.5 Year | 0.993 [0.988 to 0.996] | 0.990 [0.979 to 0.995]
  2 Years | 0.985 [0.979 to 0.990] | 0.985 [0.973 to 0.992]
  3 Years | 0.968 [0.958 to 0.975] | 0.960 [0.942 to 0.972]
  4 Years | 0.947 [0.935 to 0.956] | 0.950 [0.931 to 0.965]
  5 Years | 0.937 [0.925 to 0.948] | 0.929 [0.907 to 0.947]
  6 Years | 0.927 [0.913 to 0.938] | 0.921 [0.897 to 0.939]

12. Secondary Outcome: Percentage of Participants by Item Response to SID Satisfaction Questionnaire
Description: The SID satisfaction questionnaire was administered twice during the study and asked participants to respond to five statements using a Likert scale from "Strongly Disagree" to "Strongly Agree". Questionnaire items were as follows: "I felt comfortable injecting the study drug by myself" (Comfortable), "The SID was convenient and easy to use" (Easy to Use), "I am confident giving myself an injection in the thigh with the SID" (Confident), "Taking all things into account I find self-administration using the SID satisfactory" (Satisfactory), "If given the opportunity I would choose to continue self-injecting the study drug using the SID in the future" (Continue). Participants could only select one response per questionnaire item. There was no calculation of any score, but rather, descriptive summaries were generated by item response. The percentage of participants was reported by the response given for each item on the SID satisfaction questionnaire.
Time Frame: Cycle 4 (cycle length 3 weeks) and last safety follow-up (LSFU) (approximately 1 year)
Population: Safety Population. Only participants who performed self-administration were included. The number of participants who responded to the questionnaire item at each assessment (n) is shown in the table.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort B: SC Herceptin by SID (Self- Administered)
Number analyzed (Participants) | 550
percentage of participants
  Cycle 4: Comfortable, Strongly Disagree (n=514) | 4.7
  Cycle 4: Comfortable, Disagree (n=514) | 2.3
  Cycle 4: Comfortable, Unsure (n=514) | 7.6
  Cycle 4: Comfortable, Agree (n=514) | 41.6
  Cycle 4: Comfortable, Strongly Agree (n=514) | 43.6
  Cycle 4: Comfortable, Response Missing (n=514) | 0.2
  Cycle 4: Easy to Use, Strongly Disagree (n=514) | 3.7
  Cycle 4: Easy to Use, Disagree (n=514) | 0.6
  Cycle 4: Easy to Use, Unsure (n=514) | 1.8
  Cycle 4: Easy to Use, Agree (n=514) | 37.7
  Cycle 4: Easy to Use, Strongly Agree (n=514) | 56.0
  Cycle 4: Easy to Use, Response Missing (n=514) | 0.2
  Cycle 4: Confident, Strongly Disagree (n=514) | 3.9
  Cycle 4: Confident, Disagree (n=514) | 0.8
  Cycle 4: Confident, Unsure (n=514) | 7.2
  Cycle 4: Confident, Agree (n=514) | 42.8
  Cycle 4: Confident, Strongly Agree (n=514) | 45.1
  Cycle 4: Confident, Response Missing (n=514) | 0.2
  Cycle 4: Satisfactory, Strongly Disagree (n=514) | 3.9
  Cycle 4: Satisfactory, Disagree (n=514) | 0.6
  Cycle 4: Satisfactory, Unsure (n=514) | 2.7
  Cycle 4: Satisfactory, Agree (n=514) | 38.7
  Cycle 4: Satisfactory, Strongly Agree (n=514) | 53.9
  Cycle 4: Satisfactory, Response Missing (n=514) | 0.2
  Cycle 4: Continue, Strongly Disagree (n=514) | 3.9
  Cycle 4: Continue, Disagree (n=514) | 1.4
  Cycle 4: Continue, Unsure (n=514) | 5.3
  Cycle 4: Continue, Agree (n=514) | 33.5
  Cycle 4: Continue, Strongly Agree (n=514) | 55.8
  Cycle 4: Continue, Response Missing (n=514) | 0.2
  LSFU: Comfortable, Strongly Disagree (n=415) | 3.6
  LSFU: Comfortable, Disagree (n=415) | 3.1
  LSFU: Comfortable, Unsure (n=415) | 5.3
  LSFU: Comfortable, Agree (n=415) | 35.9
  LSFU: Comfortable, Strongly Agree (n=415) | 51.8
  LSFU: Comfortable, Response Missing (n=415) | 0.2
  LSFU: Easy to Use, Strongly Disagree (n=415) | 3.9
  LSFU: Easy to Use, Disagree (n=415) | 1.0
  LSFU: Easy to Use, Unsure (n=415) | 1.7
  LSFU: Easy to Use, Agree (n=415) | 34.9
  LSFU: Easy to Use, Strongly Agree (n=415) | 58.6
  LSFU: Easy to Use, Response Missing (n=415) | 0
  LSFU: Confident, Strongly Disagree (n=415) | 4.6
  LSFU: Confident, Disagree (n=415) | 1.2
  LSFU: Confident, Unsure (n=415) | 4.3
  LSFU: Confident, Agree (n=415) | 33.3
  LSFU: Confident, Strongly Agree (n=415) | 56.6
  LSFU: Confident, Response Missing (n=415) | 0
  LSFU: Satisfactory, Strongly Disagree (n=415) | 4.3
  LSFU: Satisfactory, Disagree (n=415) | 1.2
  LSFU: Satisfactory, Unsure (n=415) | 2.2
  LSFU: Satisfactory, Agree (n=415) | 30.8
  LSFU: Satisfactory, Strongly Agree (n=415) | 61.2
  LSFU: Satisfactory, Response Missing (n=415) | 0.2
  LSFU: Continue, Strongly Disagree (n=415) | 4.6
  LSFU: Continue, Disagree (n=415) | 1.2
  LSFU: Continue, Unsure (n=415) | 2.9
  LSFU: Continue, Agree (n=415) | 28.2
  LSFU: Continue, Strongly Agree (n=415) | 63.1
  LSFU: Continue, Response Missing (n=415) | 0

ADVERSE EVENTS:
Time Frame: Treatment Period: From Day 1 up to 19 cycles (approximately 1 year) 15 March 2015 Data Cutoff Safety Follow-up Period (SFU): From Day 1 to safety follow-up period (up to approximately 8 years)
Description: Safety Population. During the Safety Follow-up Period, no non-Serious Adverse Events occurred at the 5% frequency threshold.
  In the Safety Follow-up period, 4 participants were not included in the final analyses due to the lack of Principal Investigator signatures in the participant specific casebooks.
Groups:
- Cohort A: SC Herceptin by Needle/Syringe Safety Follow-up: Participants received SC Herceptin by an assisted administration as 600 mg every 3 weeks for a total of 18 doses/cycles. Each dose of SC Herceptin was taken from a single-use vial and injected by needle/syringe.
- Cohort B: SC Herceptin by SID Safety Follow-up: Participants received SC Herceptin as 600 mg every 3 weeks for a total of 18 doses/cycles. Each dose of SC Herceptin was administered from a pre-filled SID. The first administration was performed by an HCP. Subsequent doses were self-administered by participants who were willing and judged competent by the HCP.
Arm/Group | Cohort A: SC Herceptin by Needle/Syringe | Cohort B: SC Herceptin by SID | Cohort A: SC Herceptin by Needle/Syringe Safety Follow-up | Cohort B: SC Herceptin by SID Safety Follow-up
Serious Adverse Events (participants affected / at risk) | 242/1864 | 84/709 | 202/1862 | 53/707
Other Adverse Events (participants affected / at risk) | 1499/1864 | 576/709 | 0/1862 | 0/707
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: SC Herceptin by Needle/Syringe (N=1864) | Cohort B: SC Herceptin by SID (N=709) | Cohort A: SC Herceptin by Needle/Syringe Safety Follow-up (N=1862) | Cohort B: SC Herceptin by SID Safety Follow-up (N=707)
Neutropenic sepsis (Infections and infestations) | 9 | 1 | 0 | 0
Device related infection (Infections and infestations) | 6 | 0 | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 5 (5) | 1 | 8 (8) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 | 2 | 1 (1) | 0 (0)
Mastitis (Infections and infestations) | 3 | 2 | 4 (4) | 0 (0)
Cellulitis (Infections and infestations) | 4 | 0 | 4 (4) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 | 1 | 0 | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 4 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 2 | 1 | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 0 | 0
Breast abscess (Infections and infestations) | 2 | 0 | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 2 | 0 | 0 | 0
Infectious colitis (Infections and infestations) | 2 | 0 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 2 | 0 | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 | 1 | 0 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1 | 0 | 0
Abscess of external auditory meatus (Infections and infestations) | 1 | 0 | 0 | 0
Appendiceal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Bartholin's abscess (Infections and infestations) | 1 | 0 | 0 | 0
Breast cellulitis (Infections and infestations) | 0 | 1 | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0 | 0
Dengue fever (Infections and infestations) | 1 | 0 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 1 (1) | 0 (0)
Febrile infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 1 | 0 | 0
Hepatitis B (Infections and infestations) | 0 | 1 | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 1 | 0 | 1 (1) | 0 (0)
Intestinal sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Localised infection (Infections and infestations) | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0
Lymph node tuberculosis (Infections and infestations) | 1 | 0 | 0 | 0
Meningoencephalitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0 | 2 (2) | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0
Soft tissue infection (Infections and infestations) | 1 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0 | 0
Vaginal infection (Infections and infestations) | 1 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 1 | 2 (2) | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 39 | 14 | 1 (1) | 0
Neutropenia (Blood and lymphatic system disorders) | 9 | 6 | 0 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 3 | 0 | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Thymus enlargement (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 8 | 4 | 0 | 0
Nausea (Gastrointestinal disorders) | 5 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 3 | 0 | 1 (1) | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis erosive (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal polyp (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Subileus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 11 | 7 | 1 (1) | 1 (1)
Device breakage (Product Issues) | 1 | 1 | 1 (1) | 0 (0)
General physical health deterioration (General disorders) | 1 | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 1 (1) | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 2 (2) | 0 (0)
Death (General disorders) | 0 | 1 | 6 (6) | 1 (1)
Device defective (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 1 (1)
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 0 | 0
Non- cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 10 | 1 | 1 (1) | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 6 (6) | 0
Angina unstable (Cardiac disorders) | 2 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 2 | 0 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 2 | 0 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 1 | 0 | 0
Supraventricular tachycardia (Cardiac disorders) | 2 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 3 (3) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 1 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0 | 0
Myocarditis (Cardiac disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 1 | 0 | 0 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 0 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1 | 1 (1) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fracture displacement (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 (1) | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Traumatic arthropathy (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2 | 0 | 0
Benign pancreatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Borderline serous tumour of ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 15 (15) | 1 (1)
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 2 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 (1) | 0
Ovarian fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Schwannoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 2 (2) | 0
Syncope (Nervous system disorders) | 1 | 1 | 2 (3) | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0
Carotid sinus syndrome (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 0 | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 2 (2) | 2 (2)
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1 (2) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 (1) | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 (1) | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 4 (4) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 2 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 1 | 1 | 2 (2) | 0
Aortic aneurysm (Vascular disorders) | 1 | 0 | 0 | 0
Arterial stenosis (Vascular disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 0 | 0 | 0
Venous thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0 | 0 | 0
Ejection fraction decreased (Investigations) | 3 | 0 | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 1 | 1 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 (1) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Uterine polyp (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Breast fibrosis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Endometrial hypertrophy (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 2 (2) | 1 (1)
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 (1) | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Transient acantholytic dermatosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 2 (2) | 0 (0)
Panic attack (Psychiatric disorders) | 1 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 2 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 1 | 3 (3) | 2 (2)
Cholecystitis chronic (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 2 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 2 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0 | 1 (1) | 1 (1)
Meniere's disease (Ear and labyrinth disorders) | 1 | 0 | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 | 1 | 0 (0) | 0 (0)
Thyroiditis Subacute (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anaphylactic Shock (Immune system disorders) | 0 | 0 | 1 (1) | 1 (1)
Bile Duct Obstruction (Hepatobiliary disorders) | 0 | 0 | 1 (1) | 0 (0)
Bile Duct Stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholangitis Acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic Failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hepatic Steatosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute Hepatic Failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Renal Colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrotic Syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Bladder Polyp (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 (2) | 0 (0)
Lichen Sclerosus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 (1) | 1 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endometrial Hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 (1) | 0
Breast Necrosis (Reproductive system and breast disorders) | 0 | 0 | 1 (1) | 1 (1)
Cervical Dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1 (1) | 0
Fibrocystic Breast Disease (Reproductive system and breast disorders) | 0 | 0 | 1 (1) | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 (1) | 0
Breast Calcifications (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0
Mobility Decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0
Musculoskeletal Disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0
Scleroderma (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 (1) | 0
Thromboangiitis Obliterans (Vascular disorders) | 0 | 0 | 0 | 1 (1)
Varicose Vein (Vascular disorders) | 0 | 0 | 1 | 0
Hypertensive Urgency (Vascular disorders) | 0 | 0 | 1 (1) | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 (2) | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0
Pulmonary Sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 (1) | 0
Cerebral Infarction (Nervous system disorders) | 0 | 0 | 0 | 1 (1)
Dementia (Nervous system disorders) | 0 | 0 | 0 | 1 (1)
Dementia Alzheimer's Type (Nervous system disorders) | 0 | 0 | 0 | 1 (1)
Relapsing-Remitting Multiple Sclerosis (Nervous system disorders) | 0 | 0 | 0 | 1 (1)
Seizure (Nervous system disorders) | 0 | 0 | 0 | 1 (1)
Amyotrophic Lateral Sclerosis (Nervous system disorders) | 0 | 0 | 1 (1) | 0
Cerebral Haemorrhage (Nervous system disorders) | 0 | 0 | 1 (1) | 0
Cerebrovascular Disorder (Nervous system disorders) | 0 | 0 | 1 (1) | 0
Haemorrhagic Stroke (Nervous system disorders) | 0 | 0 | 1 (1) | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 (1) | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1 (1) | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 (1) | 0
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 (1)
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 (2) | 1 (1)
Ovarian Cancer Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 (1)
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1) | 1 (1)
Metastatic Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1) | 1 (1)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 (2) | 1 (1)
Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 (1)
Gastrointestinal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 (1)
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 (1)
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1) | 1 (1)
Lymphocytic Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1) | 0
Invasive Lobular Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1) | 0
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1) | 0
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1) | 0
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1) | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1) | 0
Endometrial Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1) | 0
Colon Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1) | 0
Chondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1) | 0
Breast Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1) | 0
Breast Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1) | 0
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1) | 0
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1) | 0
Synovial Sarcoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (2) | 0
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 3 (3) | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 2 (2)
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 (1)
Foreign Body Aspiration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 (1)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 1 (1)
Pubis Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 3 (3) | 0
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 3 (3) | 0
Clavicle Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 (2) | 0
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 (2) | 0
Rib Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 (2) | 0
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 2 (2) | 0
Intentional Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 (2) | 0
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0
Head Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0
Incisional Hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0
Post Procedural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0
Wrist Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 (1) | 0
Myocardial Infarction (Cardiac disorders) | 0 | 0 | 6 (6) | 0
Acute Coronary Syndrome (Cardiac disorders) | 0 | 0 | 1 (1) | 0
Angina Pectoris (Cardiac disorders) | 0 | 0 | 1 (1) | 0
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 | 0 | 1 (1) | 0
Atrial Flutter (Cardiac disorders) | 0 | 0 | 1 (1) | 0
Atrial Tachycardia (Cardiac disorders) | 0 | 0 | 1 (1) | 0
Cardiac Hypertrophy (Cardiac disorders) | 0 | 0 | 1 (1) | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 0 | 0 | 1 (1) | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 (1) | 0
Intracardiac Thrombus (Cardiac disorders) | 0 | 0 | 0 | 1 (1)
Sudden Death (General disorders) | 0 | 0 | 1 (1) | 0
Anal Fissure (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0
Diverticulum Intestinal (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0
Food Poisoning (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0
Hiatus Hernia (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 (1) | 0
Inguinal Hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 1 (1) | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 (1) | 0
Escherichia Sepsis (Infections and infestations) | 0 | 0 | 2 (2) | 0
Infection (Infections and infestations) | 0 | 0 | 2 (2) | 0
Biliary Tract Infection (Infections and infestations) | 0 | 0 | 1 (1) | 0
Chronic Sinusitis (Infections and infestations) | 0 | 0 | 1 (1) | 0
Dengue Haemorrhagic Fever (Infections and infestations) | 0 | 0 | 1 (1) | 0
Diabetic Gangrene (Infections and infestations) | 0 | 0 | 1 (1) | 0
Endocarditis (Infections and infestations) | 0 | 0 | 1 (1) | 0
Enterobacter Sepsis (Infections and infestations) | 0 | 0 | 1 (1) | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 0 | 1 (1) | 0
Kidney Infection (Infections and infestations) | 0 | 0 | 1 (1) | 0
Post Procedural Cellulitis (Infections and infestations) | 0 | 0 | 1 (1) | 0
Pulmonary Sepsis (Infections and infestations) | 0 | 0 | 1 (1) | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 (1) | 0
Pneumonia Influenzal (Infections and infestations) | 0 | 0 | 0 | 1 (1)
Pneumonia Streptococcal (Infections and infestations) | 0 | 0 | 0 | 1 (1)
Vulval Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1) | 0
Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1) | 0
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1) | 0
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1) | 0
Ovarian Epithelial Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1) | 0
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 (1) | 0
Keratitis (Eye disorders) | 0 | 0 | 1 (1) | 0
Anembryonic Gestation (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 (1) | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1)
Obstructive Airways Disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A: SC Herceptin by Needle/Syringe (N=1864) | Cohort B: SC Herceptin by SID (N=709) | Cohort A: SC Herceptin by Needle/Syringe Safety Follow-up (N=1862) | Cohort B: SC Herceptin by SID Safety Follow-up (N=707)
Fatigue (General disorders) | 381 | 132 | 0 | 0
Asthenia (General disorders) | 221 | 85 | 0 | 0
Pyrexia (General disorders) | 185 | 55 | 0 | 0
Oedema peripheral (General disorders) | 160 | 45 | 0 | 0
Injection site erythema (General disorders) | 128 | 52 | 0 | 0
Mucosal inflammation (General disorders) | 105 | 53 | 0 | 0
Injection site pain (General disorders) | 117 | 37 | 0 | 0
Injection site reaction (General disorders) | 101 | 36 | 0 | 0
Pain (General disorders) | 63 | 36 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 362 | 133 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 260 | 84 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 194 | 49 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 114 | 42 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 89 | 36 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 70 | 40 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 380 | 130 | 0 | 0
Nausea (Gastrointestinal disorders) | 274 | 102 | 0 | 0
Constipation (Gastrointestinal disorders) | 153 | 62 | 0 | 0
Vomiting (Gastrointestinal disorders) | 129 | 38 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 116 | 42 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 87 | 36 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 69 | 44 | 0 | 0
Headache (Nervous system disorders) | 228 | 73 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 140 | 56 | 0 | 0
Paraesthesia (Nervous system disorders) | 112 | 70 | 0 | 0
Dizziness (Nervous system disorders) | 111 | 32 | 0 (0) | 0
Peripheral sensory neuropathy (Nervous system disorders) | 94 | 21 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 177 | 74 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 156 | 74 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 163 | 49 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 115 | 35 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 190 | 56 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 115 | 47 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 109 | 30 | 0 | 0
Nasopharyngitis (Infections and infestations) | 146 | 58 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 113 | 21 | 0 | 0
Urinary tract infection (Infections and infestations) | 94 | 32 | 0 | 0
Hot flush (Vascular disorders) | 164 | 72 | 0 | 0
Hypertension (Vascular disorders) | 142 | 35 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 130 | 43 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 101 | 36 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 161 | 68 | 0 | 0
Insomnia (Psychiatric disorders) | 108 | 50 | 0 | 0
Ejection fraction decreased (Investigations) | 80 | 36 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-11-11): https://cdn.clinicaltrials.gov/large-docs/21/NCT01566721/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/21/NCT01566721/SAP_001.pdf